CLINICAL TRIAL: NCT00150930
Title: Home UVB Phototherapy for Psoriasis: Effectiveness, Quality of Life and Cost-Effectiveness
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 945-02-017; ISRCTN83025173
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2005-08

CONDITIONS: Psoriasis
Keywords: psoriasis; ultraviolet; UVB; phototherapy; home care; narrowband
MeSH Terms: conditions — Psoriasis

INTERVENTIONS:
Device: narrowband UVB phototherapy at home

SUMMARY:
UVB phototherapy is a commonly used treatment for patients with psoriasis. Generally it is performed in the outpatient department of the hospital. The UVB irradiation itself will normally take only a few minutes, but to receive the irradiation patients have to travel to the outpatient department during working hours 2 or 3 times a week. In general it is a relatively time-consuming treatment.

Objective of this study is to assess whether UVB treatment administered in the home is as equally effective as the standard outpatient UVB phototherapy. Quality of life and cost-effectiveness are also studied.

DETAILED DESCRIPTION:
Psoriasis is a chronic recurrent skin disorder characterised by erythematosquamous lesions (plaques). Usually the abnormal areas are few, but occasionally the disease is more generalised. Psoriasis can be treated locally by application of creams and ointments, for instance corticosteroids and vitamin D3. For most patients topical therapy will suffice. However, for some patients the area involved is such that topical application is not feasible. Or for others, the skin lesions do not respond anymore to topical treatment. In that case the dermatologist may start irradiation with ultraviolet (UV) light or prescribe systemic medication.

UVB phototherapy is a commonly used treatment for patients with psoriasis. Generally it is performed in the outpatient department of the hospital. The UVB irradiation itself will normally take only a few minutes, but to receive the irradiation patients have to travel to the outpatient department during working hours 2 or 3 times a week. In general it is a relatively time-consuming treatment.

To overcome the drawbacks of UVB treatment in the outpatient clinic, home UVB phototherapy was introduced over 25 years ago. However, the safety and effectiveness of home UVB have been debated ever since. Despite all discussion, the number of dermatologists prescribing home UVB phototherapy to their patients seems to gradually increase. We recently demonstrated that there is no sound evidence that would either support or dissuade from prescribing home UVB phototherapy. Particularly the lack of randomised research is apparent. Therefore, the objective of this study is to assess whether UVB treatment administered in the home is as equally effective as the standard outpatient UVB phototherapy. Quality of life and cost-effectiveness are also studied.

Primary Outcome:

(SA)PASI at inclusion, start of therapy, 23 (20-26) irradiations, end of therapy, and at every 2 months after end of therapy (maximum 1 year) Quality of life scores (EQ-5D, SF-36, PDI) at inclusion, start of therapy, 23 (20-26) irradiations and at end of therapy.

Costs and Cost-Effectiveness will be calculated with a time-horizon of 12 months after inclusion (questionnaires were used at inclusion, start of therapy, 23 (20-26) irradiations, end of therapy, and at every 2 months after end of therapy (maximum 1 year))

Secondary Outcome:

Cumulative dosimetry (every irradiation) Total amounts of and types of side-effects (every irradiation) Concomitant use of medication (during the whole trial, data derived from patients' pharmacists)

ELIGIBILITY:
Inclusion Criteria:

1. Guttate or plaque psoriasis, clinically eligible for narrowband UVB (TL-01) phototherapy;
2. Willing to undergo treatment according to randomisation.

Exclusion criteria:

1. No informed consent:

   * age below 18 years;
   * not willing to accept one of the two treatments offered;
2. Practical reasons:

   * not able to receive one of the two treatments offered (e.g. lack of space at home / living too far from hospital etc.);
   * analphabetism (unable to read the patient-information and the questionnaires, unable to provide written answers and written informed consent);
   * lack of knowledge of the Dutch language;
   * not in possession of a telephone.
3. Expected non-compliance: lack of understanding what the study / treatment is about, with its potential consequences.
4. Medical contra-indications:

   * malignancy of the skin in the past / at present;
   * known UVB-allergy or chronic polymorphic photodermatosis;
   * use (at time of inclusion) of (systemic) medication with known phototoxic or photoallergic properties;
   * use (at time of inclusion) of systemic antipsoriatic medication (cyclosporin, methotrexate, neotigason, fumaric acid);
   * history of exposure to ionising radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-10; Study Completion 2005-03

PRIMARY OUTCOMES:
(SA)PASI: whole trial (9x)
Quality of life (EQ-5D, SF-36, PDI): inclusion till end of therapy (3x)
Costs & Cost-Effectiveness: during 12 months from inclusion

SECONDARY OUTCOMES:
Dosimetry (every irradiation)
Side-effects (every irradiation)
Use medication: whole trial

CONTACTS AND LOCATIONS:
Overall Officials: Vigfús Sigurdsson, MD, PhD, Study Chair — UMC Utrecht; Mayke BG Koek, MD, M.Sc., Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Koek MB, Buskens E, Steegmans PH, van Weelden H, Bruijnzeel-Koomen CA, Sigurdsson V. UVB phototherapy in an outpatient setting or at home: a pragmatic randomised single-blind trial designed to settle the discussion. The PLUTO study. BMC Med Res Methodol. 2006 Aug 1;6:39. doi: 10.1186/1471-2288-6-39. PMID 16882343
- [Derived] Koek MB, Sigurdsson V, van Weelden H, Steegmans PH, Bruijnzeel-Koomen CA, Buskens E. Cost effectiveness of home ultraviolet B phototherapy for psoriasis: economic evaluation of a randomised controlled trial (PLUTO study). BMJ. 2010 Apr 20;340:c1490. doi: 10.1136/bmj.c1490. PMID 20406865
- [Derived] Koek MB, Buskens E, van Weelden H, Steegmans PH, Bruijnzeel-Koomen CA, Sigurdsson V. Home versus outpatient ultraviolet B phototherapy for mild to severe psoriasis: pragmatic multicentre randomised controlled non-inferiority trial (PLUTO study). BMJ. 2009 May 7;338:b1542. doi: 10.1136/bmj.b1542. PMID 19423623